CLINICAL TRIAL: NCT03863639
Title: A Pilot Study to Assess fMRI Changes and Neurocognitive Function in Women With Pre-eclampsia
Brief Title: Changes in fMRI and Neurocognitive Function in Women With Pre-eclampsia
Status: Terminated | Type: Observational
Why Stopped: Challenging enrollment
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00055293
Record Dates: First submitted 2019-03-04; First posted 2019-03-05 (Actual); Last update posted 2022-06-29 (Actual); Status verified 2022-06

CONDITIONS: Pre-Eclampsia; Neurocognitive Dysfunction
Keywords: Pre-Eclampsia; Functional Magnetic Resonance Imaging; Neurocognitive Function
MeSH Terms: conditions — Pre-Eclampsia; Cognition Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Pre-Eclampsia: 15 English-speaking women with severe pre-eclampsia
  Interventions: Diagnostic Test: Neuroimaging Procedures; Diagnostic Test: Neuropsychological Assessment Procedures
- Control: 15 English-speaking pregnant controls with uncomplicated pregnancy matched by age and gestational age
  Interventions: Diagnostic Test: Neuroimaging Procedures; Diagnostic Test: Neuropsychological Assessment Procedures

INTERVENTIONS:
Diagnostic Test: Neuroimaging Procedures — Subjects will complete neuroimaging procedures at 2-6-week postpartum or during hospitalization after delivery prior to discharge, which will consist of high-resolution anatomic, perfusion and resting-brain fMRI sequences; all of which will be acquired on a 3-Tesla General Electric magnetic resonance scanner
  provided by the Brain Imaging and Analysis Center (BIAC) at Duke University. No contrast agent will be administered in these imaging procedures.
Diagnostic Test: Neuropsychological Assessment Procedures — Once identified as meeting study criteria and consented for participation, parturients will be tested during hospitalization or as outpatients for controls, and at 2-6 weeks postpartum with the following cognitive battery. Wechsler Test of Adult Reading (WTAR), CANTABeclipse Computerized Cognitive Assessment Measures, Stroop Color-Word Test, Controlled Oral Word Association Test, EuroQol, Beck Depression Inventory Revised

SUMMARY:
This is a pilot study assessing fMRI changes and neurocognitive function in women with pre-eclampsia and healthy controls. Neurocognitive testing will be done during pregnancy and after delivery up to 2-6 weeks postpartum. fMRI will be done after delivery up to 2-6 weeks postpartum. The aims of this pilot study are therefore to 1) Determine the frequency and nature of co-morbid DTI white matter patency and fMRI functional connectivity changes in women with pre-eclampsia/eclampsia and 2) Determine the relationship between DTI white matter patency and fMRI functional connectivity changes to measurable alterations in cognitive function in this patient population. The aims of this pilot study are therefore to 1) Determine the frequency and nature of co-morbid DTI white matter patency and fMRI functional connectivity changes in women with pre-eclampsia/eclampsia and 2) Determine the relationship between DTI white matter patency and fMRI functional connectivity changes to measurable alterations in cognitive function in this patient population.

ELIGIBILITY:
Inclusion Criteria:Severe Pre-Eclampsia defined by

* Symptoms of central nervous system dysfunction (New onset cerebral or visual disturbance, such as: Photopsia, scotomata, cortical blindness, retinal vasospasm)
* Severe headache (ie, incapacitating, "the worst headache I've ever had") or headache that persists and progresses despite analgesic therapy
* Altered mental status
* Hepatic abnormality (Severe persistent right upper quadrant or epigastric pain unresponsive to medication and not accounted for by an alternative diagnosis or serum transaminase concentration ≥ twice normal, or both)
* Severe blood pressure elevation (Systolic blood pressure ≥160 mmHg or diastolic blood pressure ≥110 mmHg on two occasions at least four hours apart while the patient is on bedrest (unless the patient is on antihypertensive therapy))
* Thrombocytopenia (<100,000 platelets/microL)
* Renal abnormality (Progressive renal insufficiency (serum creatinine >1.1 mg/dL or doubling of serum creatinine concentration in the absence of other renal disease))
* Pulmonary edema

  15 English-speaking pregnant controls with uncomplicated pregnancy matched by age and gestational age will be enrolled from the antenatal clinic or the labor ward.

Exclusion Criteria:

* History of symptomatic cerebrovascular disease with substantial residual deficit
* History of alcoholism
* History of psychiatric illness
* History of claustrophobia
* Renal failure (creatinine > 2.0 mg/dl)
* Patients with less than a 7th grade education or unable to read and thus unable complete the neuropsychological testing
* Patients with bodily implants unsafe for MRI use

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Parturients with severe pre-eclampsia on the labor and delivery ward and healthy controls presenting to the antenatal clinic or the labor ward will be screened. 15 English-speaking pregnant controls with uncomplicated pregnancy matched by age and gestational age will be enrolled from the antenatal clinic or the labor ward.
Sampling Method: Non-Probability Sample
Enrollment: 18 (Actual)
Dates: Start 2014-07-07 (Actual); Primary Completion 2022-04-13 (Actual); Study Completion 2022-04-13 (Actual)

PRIMARY OUTCOMES:
Number of white matter lesions | Postpartum (2-6 weeks or while hospitalized)
  DTI white matter patency in women with pre-eclampsia/eclampsia.
Classification of white matter lesions | Postpartum (2-6 weeks or while hospitalized)
  Classify the nature of co-morbid DTI white matter patency/lesions
Neurocognitive Function Scores | Up to 1 day before delivery
  Scores from the neurocognitive testing combined to give overall score for function.

CONTACTS AND LOCATIONS:
Overall Officials: Ashraf S Habib, MD, Principal Investigator — Duke University
Locations (1):
- Duke University Medical Center, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No